CLINICAL TRIAL: NCT01858883
Title: Official Title: A Phase 1B/2 Study of the Safety and Tolerability of Itacitinib (INCB039110) in Combination With Gemcitabine and Nab-Paclitaxel in Subjects With Advanced Solid Tumors
Brief Title: Safety Study of Itacitinib (INCB039110) in Combination With Gemcitabine and Nab-Paclitaxel in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 39110-116
Record Dates: First submitted 2013-05-14; First posted 2013-05-21 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Solid Tumors; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — itacitinib; INCB039110; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- itacitinib, gemcitabine, nab-paclitaxel, filgrastim (Experimental)
  Interventions: Drug: itacitinib; Drug: Gemcitabine; Drug: nab-paclitaxel; Drug: filgrastim

INTERVENTIONS:
Drug: itacitinib
  Other Names: INCB039110
Drug: Gemcitabine
  Other Names: Gemzar®
Drug: nab-paclitaxel
  Other Names: Abraxane®
Drug: filgrastim
  Other Names: Neupogen®

SUMMARY:
Test the hypothesis that itacitinib (INCB039110) can be administered safely in combination with gemcitabine and nab-paclitaxel in subjects with advanced or metastatic cancer.

DETAILED DESCRIPTION:
Study Part 1: This is a dose optimization phase designed to find a tolerated regimen that includes identifying the MTD of itacitinib (INCB039110) (within a defined pharmacologic range) in combination with doses of gemcitabine and nab-paclitaxel that have established safety and tolerability in subjects with advanced or metastatic solid tumors.

Study Part 2 and Part 2A: This phase will explore the safety and tolerability of the MTD or PAD of itacitinib (INCB039110) when administered in combination with gemcitabine and nab-paclitaxel in subjects with untreated advanced or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor (Part 1) or pancreatic adenocarcinoma (Part 2)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Received no more than 1 prior chemotherapy regimen for advanced or metastatic disease (not including neo-adjuvant and/or adjuvant therapy) (Part 1)
* Received no prior chemotherapy for advanced or metastatic disease (Part 2 and Part 2a)
* Adequate renal, hepatic, and bone marrow function without frequent blood product or hematopoietic growth factor support (eg use of erythropoietin or transfusions > 2 units packed red blood cells every 3 months)
* Ability to swallow and retain oral medication

Exclusion Criteria:

* Any known contraindications to the use of a required comedication (gemcitabine or nab-paclitaxel).
* Evidence of uncontrolled brain metastases or history of uncontrolled seizures.
* Ongoing radiation therapy and/or radiation therapy administered within 28 days of enrollment or ongoing radiotherapy-related toxicities.
* Presence of ≥ Grade 2 neuropathy.
* Inability to swallow food or any condition of the upper GI tract that precludes administration of oral medications.
* Recent (≤ 3 months) history of partial or complete bowel obstruction.
* Unwillingness to be transfused with blood components.
* Known history of Hepatitis B or C infection or HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-06; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of combination therapy study treatment itacitinib (INCB039110) plus nab-paclitaxel and gemcitabine as measured by the number of participants with adverse events | Baseline and weekly for Cycle 1 and then Day 1, Week 8 and Week 15 for all subsequent cycles until the End of Treatment visit (approximately 6 months).
Identify the Maximum Tolerated Dose (MTD) or Pharmacologically Active Dose (PAD) within a defined dose range for itacitinib (INCB039110) in the treatment regimens administered | Each cohort will be observed for a minimum of 28 days.

SECONDARY OUTCOMES:
Pharmacokinetics of gemcitabine and paclitaxel administered with or without concurrent itacitinib (INCB039110) | Baseline up to 6 months.
Clinical activity as measured by the greatest decrease in tumor burden compared to baseline. | Baseline and approximately every two cycles throughout the study until study completion or early termination (approximately 6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Albert Assad, M.D., Study Director — Incyte Corporation
Locations (8):
- United States (8):
  - Scottsdale, Arizona
  - Fayetteville, Arkansas
  - Beverly Hills, California
  - Southington, Connecticut
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Lake Success, New York
  - Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Beatty GL, Shahda S, Beck T, Uppal N, Cohen SJ, Donehower R, Gabayan AE, Assad A, Switzky J, Zhen H, Von Hoff DD. A Phase Ib/II Study of the JAK1 Inhibitor, Itacitinib, plus nab-Paclitaxel and Gemcitabine in Advanced Solid Tumors. Oncologist. 2019 Jan;24(1):14-e10. doi: 10.1634/theoncologist.2017-0665. Epub 2018 Aug 16. PMID 30115734